CLINICAL TRIAL: NCT05204303
Title: Analysis of Mouthwash Samples From Laryngopharyngeal Reflux (LPR) Patients and Healthy Volunteers Using Barrel-array Diagnostics
Brief Title: LPR Fluorescence Pilot
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Functional Gut Clinic (Other)
Collaborators: Rosa Biotech (Unknown)
Responsible Party: Principal Investigator, Dr Anthony Hobson, Clinical Director, The Functional Gut Clinic
Other Study IDs: FGC-22-001
Record Dates: First submitted 2022-01-10; First posted 2022-01-24 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: Laryngopharyngeal Reflux; Gastro Esophageal Reflux
MeSH Terms: conditions — Laryngopharyngeal Reflux; Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Mouthwash (salivary oral rinse)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with symptoms of LPR and objective evidence of GORD
  Interventions: Diagnostic Test: 24-hour pH-impedance monitoring; Other: Symptom questionnaires; Other: ROME IV Diagnostic Questionnaire
- Patients with symptoms of LPR and no objective evidence of GORD
  Interventions: Diagnostic Test: 24-hour pH-impedance monitoring; Other: Symptom questionnaires; Other: ROME IV Diagnostic Questionnaire
- Healthy volunteers
  Interventions: Other: Symptom questionnaires; Other: ROME IV Diagnostic Questionnaire

INTERVENTIONS:
Diagnostic Test: 24-hour pH-impedance monitoring — Ambulatory transnasal reflux device to detect reflux events in the oeosphagus and pharynx.
  Groups: Patients with symptoms of LPR and no objective evidence of GORD; Patients with symptoms of LPR and objective evidence of GORD
Other: Symptom questionnaires — Reflux Symptom Index (RSI) Gastroesophageal Reflux Disease Questionnaire (GERDQ) Short-form Esophageal Hypervigilance and Anxiety Scale (SF-EHAS)
Other: ROME IV Diagnostic Questionnaire — A symptom-based questionnaire used to diagnose disorders of gut-brain interaction (DGBI)

SUMMARY:
Comparing the fluorescence signatures from mouthwash samples of patients with laryngopharyngeal reflux (LPR) and healthy volunteers.

DETAILED DESCRIPTION:
The investigators aim to test if the biosensing platform Pandra, developed by Rosa Biotech, may be suitable to distinguish patients with LPR symptoms, both with and without objective evidence of gastroesophageal reflux disease (GORD), vs healthy volunteers due to their expected inflammation and cell changes in the laryngo-pharyngeal region. The investigators intend to analyse 20 samples of mouthwash solutions from each of the following groups:

A. Patients with symptoms of LPR and objective evidence of GORD B. Patients with symptoms of LPR and no objective evidence of GORD C. Healthy volunteer group

ELIGIBILITY:
Healthy Volunteers

Inclusion Criteria:

* Participant is Aged 18 or above
* Participant has capacity to understand written English
* Participant is not on regular prescription medicines
* Participant has an RSI score of 0
* Participant has a body mass index (BMI) of 18.5 - 34.9 kg/m2 (bounds included)

Exclusion Criteria:

* Participant has experienced any symptoms of LPR or GORD symptoms in the past year
* Participant has taken any medication for GORD/LPR in the past year (e.g. proton pump inhibitors, h2 antagonists, over the counter antacids)
* Participant has active oral disease
* Participant has a significant medical diagnosis

Patients with symptoms of LPR

Inclusion Criteria:

* Participant is Aged 18 or above
* Participant has capacity to understand written English
* Participant has an RSI score of >13
* Participant has a body mass index (BMI) of 18.5 - 34.9 kg/m2 (bounds included
* Participant has been referred for 24hr ambulatory pH-impedance monitoring

Exclusion Criteria:

* Participant has active oral disease
* Participant has other ongoing health problems that could account for their LPR symptoms.
* Participant has NOT undergone nasoendoscopy within last 6 months OR does not have one scheduled within next 6 weeks
* Previous antireflux surgery (e.g. fundoplication or magnetic sphincter augmentation)
* Previous bariatric surgery (e.g. gastric bypass or sleeve gastrectomy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with LPR symptoms referred for ambulatory pH-impedance monitoring will be separated into two groups following completion of the pH-impedance test: those with objective evidence of GORD and those without objective evidence of GORD.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Determine the detection strength of differences in fingerprints between the three participant groups. | 10-months

SECONDARY OUTCOMES:
Determine the differences in fingerprints between samples within one group to assess background noise. | 10-months
Determine the feasibility of mouthwash on Pandra platform. | 10-months

CONTACTS AND LOCATIONS:
Locations (1):
- The Functional Gut Clinic, Manchester, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No